CLINICAL TRIAL: NCT02820727
Title: Perioperative Three Dimensional Right Ventricular Function
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AnTubingen-RV
Record Dates: First submitted 2016-06-06; First posted 2016-07-01 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2016-06

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study addresses the influence of anesthesia induction, ventilation and influence of cardiac surgical procedures and cardio-pulmonary-bypass on right ventricular function. Influence on patient outcome is also studied. Three dimensional echocardiography is applied.

ELIGIBILITY:
Inclusion Criteria:

* informed consent given
* cardiac surgical procedure
* left sided cardiac surgery or bypass surgery, ascending aortic surgery, assist device implantation

Exclusion Criteria:

* pregnant patients
* contraindication for transesophageal echocardiography

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Time on Intensive Care Unit (ICU) | up to 60 days
  Duration of ICU stay

SECONDARY OUTCOMES:
Time to hospital discharge | up to 120 days
  Hospital Outcome
Catecholamine dosages | up to 24 hours
  after anesthesia induction, end of surgery, 12h and 24h after intensive care unit (ICU) admission
Catecholamine free days | up to 60 days
  Catecholamine free days on ICU
Hours on mechanical ventilation | up to 1440 hours
  Duration of mechanical ventilation
Organ failure during ICU stay | up to 60 days
  Early organ failure (Lab tests: Creatinine, Bilirubin, Lactate, Thromboplastin Time)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Magunia, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tubingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Magunia H, Jordanow A, Keller M, Rosenberger P, Nowak-Machen M. The effects of anesthesia induction and positive pressure ventilation on right-ventricular function: an echocardiography-based prospective observational study. BMC Anesthesiol. 2019 Nov 4;19(1):199. doi: 10.1186/s12871-019-0870-z. PMID 31684877